CLINICAL TRIAL: NCT04331418
Title: Comparison of Caudal Block Versus Dexmedetomidine Infusion in Pediatric Patients Undergoing Hypospadias Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Faheem, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: precedex infusion in pediatric
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Dexmedetomidine Infusion; Pediatric; Hypospadias Repair Surgery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): On arrival to operating room, Noninvasive monitors, such as electrocardiography, noninvasive blood pressure (NIBP), oxygen saturation (SpO2), will be attached and baseline parameters such as heart rate, mean arterial pressure, and peripheral oxygen saturation will be recorded .
  General anesthesia will be induced with O2/sevo (FiO2 = 1 /sevoflurane 8% MAC), cis-atracurium 0.1 mg/kg iv, +/- fentanyl 1 mcg/kg iv. Trachea will be intubated with an appropriate sized, endotracheal tube and maintenance of anesthesia by O2/Air (FiO2 = 0.4), sevoflurane 2% MAC.
  Dexamethasone 0.15 mg/kg iv will be given as PONV prophylaxis. Increments of fentanyl 0.5 mcg/kg iv and cis-atracurium 0.03 mg/kg iv will be given according to hemodynamics and capnography.
- caudal group (Experimental): After negative aspiration of blood or cerebrospinal fluid, 2 mg/ kg of bupivacaine at concentration of 0.5% (volume 0.5ml/kg) was given as per the group assigned, then the site of injection was dressed, and the patient was turned supine.
  Interventions: Procedure: caudal block
- dexmetomidine group (Experimental): Children in this group will be received (1 mcg/kg IV over 10 minutes followed by 0.5 mcg/kg/hr) with a suggested maximum dose of 2 mcg/kg.of dexmedetomidine is available in a 100 mcg/mL concentration in a 2 mL preservative-free vial. It may be prepared as a 2 to 4 mcg/mL solution using normal saline
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 1 mcg/kg IV over 10 minutes followed by 0.5 mcg/kg/hr
  Arms: dexmetomidine group
Procedure: caudal block — After negative aspiration of blood or cerebrospinal fluid, 2 mg/ kg of bupivacaine at concentration of 0.5% (volume 0.5ml/kg) was given as per the group assigned, then the site of injection was dressed, and the patient was turned supine.
  Arms: caudal group

SUMMARY:
Pain is one of the most misunderstood, underdiagnosed, and untreated medical problems, particularly in children. New Joint Commission on Accreditation of Health Care Organization regards pain as fifth vital sign and requires caregivers to regularly assess pain. Inadequate pain relief during childhood may have long-term negative effects including harmful neuroendocrine responses disrupted eating and sleep cycles and increased pain perception during subsequent painful experiences. Also, postoperative pain can result in an uncooperative and restless child. Hence, it is preferable to prevent the onset of pain rather than to relieve its existence.

Various multimodal techniques have been designed for pediatric pain relief. These include both systemic and regional analgesia. The most commonly used regional technique is caudal epidural block. Advantages of the caudal block are smoother recovery with less distress behavior, early ambulation, decreased the risk of chest infections, decreased postoperative analgesic requirements, and early discharge.

In our culture; considerable number of parents still refuses caudal anesthesia fearing from the rare neurological sequelae may occur. This the motive for searching for parenteral surrogate gives clear headed recovery resembles regional analgesia.

Dexmedetomidine is an alpha 2 agonist which has sedative, analgesic, and opioid-sparing effect. It prolongs the duration of analgesia by its local vasoconstrictive effect and by increasing the potassium conductance in A-delta and C-fibers.

It also exerts its analgesic action centrally via systemic absorption or by diffusion into the cerebrospinal fluid and reaches alpha 2 receptors in the superficial laminae of the spinal cord and brainstem or indirectly activating spinal cholinergic neurons. The sedative effects of dexmedetomidine are mostly due to stimulation of the alpha 2 adrenoceptor in the locus coeruleus

ELIGIBILITY:
Inclusion Criteria:

1. male children
2. american society of aneasthesia physical status grade I &II
3. patients aged from 2 years to 12 years
4. patients will undergoing hypospadias repair surgery

Exclusion Criteria:

1. history or evidence of infection at the back
2. allergy to the study drugs
3. bleeding/coagulation disorder
4. developmental delay
5. septic patients
6. neurological or spinal diseases.

Ages: 2 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 135 (Actual)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
quality of recovery of the studied patients | in immediate recovery from aneasthesia at postaneathetic care unit up to 2 hours
  quality of recovery of the studied patients using modified objective pain score
quality of recovery of the studied patients | from discharge from PACU up to 6 hours in the surgical ward
  change in quality of recovery of the studied patients using modified objective pain score

SECONDARY OUTCOMES:
concentration of required postoperative analgesic | in immediate recovery from aneasthesia up to 2 hours at postaneathetic care unit
  concentration of postoperative analgesic
concentration of required postoperative analgesic | from discharge from PACU up to 6 hours in the surgical ward
  concentration of required postoperative analgesic
concentration of required postoperative sedation | in immediate recovery from aneasthesia up to 2 hours at postaneathetic care unit
  concentration of required postoperative sedation
concentration of required postoperative sedation | from discharge from PACU up to 6 hours in the surgical ward
  concentration of required postoperative sedation
number of patients developed perioperative complications. | in immediate recovery from aneasthesia up to 2 hours at postaneathetic care unit
  number of patients developed perioperative complications
number of patients developed perioperative complications. | from discharge from PACU up to 6 hours in the surgical ward
  number of patients developed perioperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdelrahman, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No